CLINICAL TRIAL: NCT03167502
Title: Performance in Walking in Osteoarthritis Patients: the Role of Fatigue and the Effect of an Eccentric Muscle Building Program
Brief Title: Performance in Walking in Osteoarthritis Patients
Acronym: EX-ART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16-AOIP-03
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- concentric work (Active Comparator): patient suffering from knee osteoarthritis will follow a concentric work. This training is 2 sessions per week for 6 weeks
  Interventions: Other: concentric work
- eccentric work (Experimental): patient suffering from knee osteoarthritis will follow an eccentric work. This training is 2 sessions per week for 6 weeks
  Interventions: Other: eccentric work

INTERVENTIONS:
Other: eccentric work — patient will follow 2 eccentric trainings per week during 6 weeks
  Arms: eccentric work
Other: concentric work — patient will follow 2 concentric trainings per week during 6 weeks
  Arms: concentric work

SUMMARY:
Few data exist to date on the effect of eccentric muscle building in knee osteoarthritis. No studies have compared the effect of eccentric versus concentric reinforcement in knee osteoarthritis. Our study aims to show the effectiveness of an eccentric reinforcement. This is a randomized, interventional trial.

DETAILED DESCRIPTION:
Few data exist to date on the effect of eccentric muscle building in knee osteoarthritis. No studies have compared the effect of eccentric versus concentric reinforcement in knee osteoarthritis. Our study aims to show the effectiveness of an eccentric reinforcement, the interest of a work supervised by a sports coach to maintain activity over time and to study the effect of this activity at the muscular level. The main objective is to study the effect of an eccentric muscle strengthening program on walking performance in osteoarthritis patients. The secondary objectives are to study: the effect of fatigue on walking, the relationship between fatigue and the level of physical activity, the effect of training on perceived fatigue and the effect of training on the function and at muscular level. This is a randomized, interventional trial. 40 subjects are planned. Inclusion criteria include: age 40-85 years, KL 2 and 3. The subjects are divided into two groups to perform either eccentric or concentric work. 2 sessions per week for 6 weeks. At baseline and at the end of the study a clinical evaluation and MRI will be carried out for evaluation of the criteria of judgment

ELIGIBILITY:
Inclusion Criteria:

* Autonomous subjects aged 40 to 85
* Subjects meeting ACR criteria for gonarthrosis
* Subjects with a score of Kellgren and Lawrence at least one knee greater than or equal to 2
* Signature of consent form
* Subjects affiliated to social security

Exclusion Criteria:

Subject with a Kellgren and Lawrence stadium at 4 for at least one of his two knees

* Subjects with symptomatic femoro-patellar arthrosis
* Subject with a pathology that makes walking testing impossible.
* Non-autonomous subjects, with a pathology impairing walking
* Subjects with symptomatic osteoarthritis of the hip and / or with a hip or knee prosthesis
* Subject incapable of signing consent and unable to understand information leaflet.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2017-11-25 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
Walking performance | after 6 training weeks
  6-minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Christian H ROUX, PhD, Principal Investigator — service de Rhumatologie, CHU de NICE
Locations (1):
- Department of rheumatology, nice university hospital, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Trojani MC, Chorin F, Gerus P, Breuil V, Michel C, Guis S, Bendahan D, Roux C. Concentric or eccentric physical activity for patients with symptomatic osteoarthritis of the knee: a randomized prospective study. Ther Adv Musculoskelet Dis. 2022 Jul 7;14:1759720X221102805. doi: 10.1177/1759720X221102805. eCollection 2022. PMID 35832351